CLINICAL TRIAL: NCT02159339
Title: A Cohort Study on Prediction of Metastasis of Gastric Carcinoma by DNA Methylation Biomarkers
Brief Title: DNA Methylation Biomarkers and Metastasis of Gastric Carcinoma
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Zhaojun Liu, Zhaojun Liu, Peking University Cancer Hospital & Institute
Other Study IDs: Methylation-14414
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Gastric Carcinoma
Keywords: DNA methylation
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue specimens are surgically collected from inpatients with pN0M0-stage gastric carcinoma. Genomic DNA sample is extracted from tissues. Unmethylated cytosine residues in DNA are converted into uracil residues with bisulfite modification.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- gene-methylation: gene-low-level of methylation: patients with early stage gastric carcinoma containing low-level of methylation change of E-cadherin,GFRA1,p16,SRF and ZNF382 CpG island.
  gene-middle-level of methylation: patients with early stage gastric carcinoma containing middle-level of methylation change of E-cadherin,GFRA1,p16,SRF and ZNF382 CpG island.
  gene-high-level of methylation: patients with early stage gastric carcinoma containing high-level of methylation change of E-cadherin,GFRA1,p16,SRF and ZNF382 CpG island.
  gene-without of methylation: patients with early stage gastric carcinoma NOT containing methylated E-cadherin,GFRA1,p16,SRF or ZNF382 CpG island.

SUMMARY:
Gastric carcinoma (GC) is the second leading cause of cancer death throughout the world. In previous multi-center study, we have found that the prevalence of GDNF family receptor alpha 1(GFRA1), serum response factor (SRF), and ZNF382 methylation alterations were inversely and coordinately associated with GC metastasis and the patients' overall survival throughout discovery and testing cohorts in China, Japan and Korea. The present cohort study is to investigate whether methylation of those genes can predict the metastasis and prognosis of GC.

DETAILED DESCRIPTION:
Background: Metastasis is the leading cause of death for gastric carcinoma (GC). Currently, GC prognosis is primarily determined based on the clinical data and pathological stages of patients at the time of diagnosis and treatment. However, successful management of GC patients is still hampered by lack of highly sensitive and specific biomarkers capable of predicting prognosis and likelihood of metastasis. GFRA1 hypomethylation along with SRF and ZNF382 hypermethylation were found to be potential synergistic biomarkers for the prediction of GC metastasis in our previous multi-center study. In addition, p16 and E-cadherin were also correlated with GC metastasis in Chinese cohort. To investigate the predictive value of those genes' methylation on metastasis potential in GC, we carried out the prospective cohort study.

Methods: 198 early stage GC patients without lymph node or distal metastasis were included in the present study. Baseline information of E-cadherin, GFRA1, p16, SRF and ZNF382 methylation status of the GC from 191 cases was obtained by MethyLight. The follow-up examination was carried out in a double-blind study with a 6-month interval. The association between gene methylation and metastasis of GC was analyzed with SPSS16.0 software. All P-values were two-sided.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of gastric adenocarcinoma;
* Early stage GC without lymph node and distal metastasis;
* Availability of frozen, fresh GC and corresponding surgical margin samples;
* Available of methylation status of gene CpG island in the extracted DNA sample.

Exclusion Criteria:

* GC with lymph node or distal metastasis;
* Quality of the prepared DNA is not good enough for detection of gene methylation;
* GC cases were subjected to the neoadjuvant chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 198 early stage gastric carcinoma (GC) inpatients that underwent surgical treatment at Peking University Cancer Hospital & Institute between 2002 and 2012 were enrolled in the cohort. All of the enrolled patients had been diagnosed pathologically by senior pathologists. The 2010 UICC-TNM (tumor-node-metastasis) system was used for the classification of GCs. All cases involved primary lesions without neoadjuvant chemotherapy. Genes methylation status of GC samples was analyzed with MethyLight combined with denatured high performance liquid chromatography. 191 eligible cases with gene-methylated or gene-methylated GC were enrolled into the cohort study.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Metastasis and/ or recurrence of gastric carcinoma | 3 years
  The hazard ratio, positive prediction value, and negative prediction value of metastasis/recurrence of gastric carcinomas are calculated according to the metastasis/recurrence frequences among patients with the different methylation status of each target gene CpG islands. These patients are classified into four groups for each gene: A) cases without methylation change; B) cases with the low-level of methylation change (33.3% of cases with methylation change); C) cases with the middle-level of methylation change (33.3% of cases with methylation change); D) cases with the high-level of methylation change (33.3% of cases with methylation change). Combination analysis will be carried out using Support Vector Classification model.

SECONDARY OUTCOMES:
Disease-free (Recurrence/metastasis-free) survival (DFS) and overall survival (OS) of patients with gastric carcinoma after surgical resection | from 4 months to 144 months
  The classification of patients is the same as the primary outcome measure. The log-rank test will be used to compare survival time between groups. Cox-proportional hazards models will be used to identify independent predictors of survival (month) with adjustment for relevant clinical covariates

CONTACTS AND LOCATIONS:
Overall Officials: Dajun Deng, Master, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital & Institute, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Cao J, Zhou J, Gao Y, Gu L, Meng H, Liu H, Deng D. Methylation of p16 CpG island associated with malignant progression of oral epithelial dysplasia: a prospective cohort study. Clin Cancer Res. 2009 Aug 15;15(16):5178-83. doi: 10.1158/1078-0432.CCR-09-0580. Epub 2009 Aug 11. PMID 19671846
- [Derived] Liu Z, Cheng X, Zhang L, Zhou J, Deng D, Ji J. A panel of DNA methylated markers predicts metastasis of pN0M0 gastric carcinoma: a prospective cohort study. Br J Cancer. 2019 Oct;121(7):529-536. doi: 10.1038/s41416-019-0552-0. Epub 2019 Aug 21. PMID 31431673